CLINICAL TRIAL: NCT06712498
Title: INVESTIGATION OF THE INTRAOPERATIVE AND POSTOPERATIVE EFFECTS
Brief Title: INVESTIGATION OF THE INTRAOPERATIVE AND POSTOPERATIVE EFFECTS OF EXTERNAL OBLIQUE INTERCOSTAL PLAN BLOCK IN PATIENTS UNDERGOING LAPARASCOPIC CHOLESYSTECTOMY OPERATION
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mazlum Dursun, Anesthesiology and Reanimation spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: mazlum
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-11

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- External oblique intercostal plan block group: After endotracheal intubation, a 22-gauge 100 mm long block needle will be inserted at the T6-T7 level under USG guidance and bilateral EOIB will be applied with 20 cc of 0.25% Bupivacaine on each side under the external oblique intercostal muscle (total 40ml bilaterally).
  Interventions: Procedure: External Oblique Intercostal Plane Block
- control group: No Intervention
  Interventions: Drug: control group

INTERVENTIONS:
Procedure: External Oblique Intercostal Plane Block — After endotracheal intubation, a 22-gauge 100 mm long block needle will be inserted at the T6-T7 level under USG guidance and bilateral EOIB will be applied with 20 cc of 0.25% Bupivacaine on each side under the external oblique intercostal muscle (total 40ml bilaterally).
  Groups: External oblique intercostal plan block group
Drug: control group — No intervention
  Groups: control group

SUMMARY:
Objective: Regional anesthesia techniques, such as peripheral nerve blocks, have a lower side effect profile and higher patient satisfaction compared to central blocks. With the introduction of Ultrasonography (USG), these techniques have become more commonly and reliably performed. The purpose of our study is to compare parameters such as intraoperative hemodynamics, postoperative analgesic requirement, and patient satisfaction between patients undergoing External Oblique Intercostal Plane Block (EOIB) with those who did not receive EOIB, which has few studies conducted on it.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-65
* and with ASA1-2 were included.

Exclusion Criteria:• Patients younger than 18 years of age and older than 65 years of age

* Patients allergic to local anesthetics
* Patients with opioid and alcohol addiction
* Patients with perioperative signs of acute cholecystitis
* Patients with contraindications for laparoscopic surgery
* Cases with ASA III-IV were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: operating
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Postoperative 30.second,2 hours, 6 hours,12 hours,24 hours
  They will be numbered from 1 to 10. If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome
Visual Analogue Scale | Postoperative 30.second,2 hours, 6 hours,12 hours,24 hours
  The Visual Analogue Scale (VAS) is a subjective measure of pain. It consists of a 10cm line with two endpoints representing 'no pain' and 'worst pain imaginable'. Patients are asked to rate their pain by placing a mark on the line corresponding to their current level of pain. The distance along the line from the 'no pain' marker is then measured with a ruler giving a pain score out of 10.

SECONDARY OUTCOMES:
Riker Sedation Agitation Scale | Immediately after extubation
  7 Dangerous Agitation ... If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Patient satisfaction score | at the 24th postoperative hour
  Patients' satisfaction with the quality of pain management will be evaluated on the second postoperative day using the following scale: 1 = very unsatisfied; 2 = highly dissatisfied; 3 = medium; 4 = very satisfactory; 5 = very satisfactory
Postoperative vomiting and nausea | Postoperative 30.second,2 hours, 6 hours,12 hours,24 hours
  Postoperative vomiting and nausea: yes or no
Opioid use | Postoperative 24 hours
  Tramadol use
Mean Arter Pressure | when you come to the operating room table, after block Intraoperative 10 minutes,30 minutes postoperative 2,6,12 hours
  mm/hg
Heart Rate | when you come to the operating room table, after block Intraoperative 10 minutes,30 minutes postoperative 2,6,12 hours
  beats/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Diyarbakır, Kayapınar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No